CLINICAL TRIAL: NCT02689882
Title: "Pharmacokinetic Study of Nicotinamide Riboside"
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kevin O'Brien, Professor of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HL126209-01S1; R21HL126209-01S1 (NIH)
Record Dates: First submitted 2016-02-16; First posted 2016-02-24 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Metabolic Disturbance
Keywords: nicotinamide riboside; nicotinamide ribonucleoside; Nicotinamide-Adenine Dinucleotide
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pharmacokinetic study (Experimental): Nicotinamide riboside dose up-titration: Days 1 and 2: 250 mg by mouth daily; Days 3 and 4: 250 mg by mouth twice daily; Days 5 and 6: 500 mg by mouth twice daily; Days 7 and 8: 1000mg by mouth twice daily; Day 9: single dose of 1000mg by mouth followed by 24 hour pharmacokinetic study.
  Interventions: Dietary Supplement: nicotinamide riboside

INTERVENTIONS:
Dietary Supplement: nicotinamide riboside — Nicotinamide riboside dose up-titration: Days 1 and 2: 250 mg by mouth daily; Days 3 and 4: 250 mg by mouth twice daily; Days 5 and 6: 500 mg by mouth twice daily; Days 7 and 8: 1000mg by mouth twice daily; Day 9: single dose of 1000mg by mouth followed by 24 hour pharmacokinetic study.
  Other Names: Niagen

SUMMARY:
Nicotinamide riboside (NR) has been available over the counter as a nutraceutical (Niagen®, ChromaDex, Inc.) since the summer of 2013. However, classical pharmacokinetic (PK) data for NR have not been reported in humans. This study will use a recently-developed, whole blood assay for NR to assess the pharmacokinetics of NR at a maximum dose of 1000 mg twice daily, and will collect history, physical examination and laboratory data to determine the safety and tolerability of NR in eight, healthy volunteers. In addition, whole blood nicotinamide adenine dinucleotide (NAD) levels will be measured at each time point, to determine whether this NR dose significantly raises whole blood NAD levels.

DETAILED DESCRIPTION:
1. On Day 1, participants will have a baseline assessment, including blood pressure and heart rate, as well as baseline assessment of "safety" labs: complete blood count with white blood count differential and platelets, serum chemistry panel (sodium, potassium, chloride, glucose, blood urea nitrogen and creatinine), uric acid, creatine kinase, aspartate aminotransferase and alanine aminotransferase, and lactate dehydrogenase.
2. Participants will receive 250 mg nicotinamide riboside (NR) by mouth daily on Days 1-2, 250 mg NR by mouth twice daily on Days 3-4, 500 mg NR twice daily by mouth on Days 5-6 and 1000 mg NR twice daily by mouth on Days 7-8.
3. On Day 2, a blood sample will be obtained from each participant to measure serum chemistry panel to assess for the possibility of hyperkalemia and hyperglycemia. In addition, an instant read potassium will be measured using a point-of-care device available on the University of Washington (UW) General Clinical Research Center (GCRC). If the potassium is greater than 5.5, a repeat value and an ECG will be performed and the Study Investigator. If it is greater than 6.0, the Study Investigator will evaluate the subject for admission.
4. On Day 9 prior to receiving their morning dose, participants will be admitted to the UW GCRC for an overnight stay.

   1. In the UW GCRC, the participants will receive the last 1000 mg dose of NR at time=0.
   2. Blood samples will be collected at time = 30 minutes and at 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours.
   3. Whole blood samples will be frozen at -80 degrees C until assayed for NR and NAD+.
   4. "Safety labs" performed on Day 1 will be repeated

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult (age 21-50 years), male or female
* Willing and able to provide informed consent

Exclusion Criteria:

* Current smoking
* Receiving concurrent medications or supplements
* History of liver, renal, cardiovascular, endocrine, or neurological disease
* Known allergy to niacin or nicotinamide ribosome
* Unwilling to refrain from drinking alcohol during the duration of the study

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percent change in the average steady state concentration (Css) of nicotinamide riboside (NR) on day 9 (following up titration of nicotinamide riboside to 1000 mg by mouth twice daily) compared to pre-dose baseline. | 9 days
  Percent change in the average steady state concentration (Css) of nicotinamide riboside (NR) on day 9 (following up titration of nicotinamide riboside to 1000 mg by mouth twice daily) compared to pre-dose baseline. Group mean values will be compared by paired t-test, with correction for multiple primary endpoints.
Percent change in the average steady state concentration (Css) of nicotinamide adenine dinucleotide (NAD) on day 9 (following up titration of nicotinamide riboside to 1000 mg by mouth twice daily) compared to pre-dose baseline. | 9 days
  Percent change in the average steady state concentration (Css) of nicotinamide adenine dinucleotide (NAD) on day 9 (following up titration of nicotinamide riboside to 1000 mg by mouth twice daily) compared to pre-dose baseline. Group mean values will be compared by paired t-test, with correction for multiple primary endpoints.

SECONDARY OUTCOMES:
Effect of nicotinamide riboside on serum potassium levels | 9 days
  Comparison of group mean serum potassium levels at day 1 (baseline) vs. day 9 (while on nicotinamide riboside 1000mg twice daily). Group mean potassium levels will be compared by paired t-test, with correction for multiple comparisons.
Effect of nicotinamide riboside on serum creatine kinase levels | 9 days
  Comparison of group mean serum creatine kinase levels at day 1 (baseline) vs. day 9 (while on nicotinamide riboside 1000mg twice daily). Group mean creatine kinase levels will be compared by paired t-test, with correction for multiple comparisons.
Effect of nicotinamide riboside on serum glucose levels | 9 days
  Comparison of group mean serum glucose levels at day 1 (baseline) vs. day 9 (while on nicotinamide riboside 1000mg twice daily). Group mean glucose levels will be compared by paired t-test, with correction for multiple comparisons.
Effect of nicotinamide riboside on serum uric acid levels | 9 days
  Comparison of group mean serum uric acid levels at day 1 (baseline) vs. day 9 (while on nicotinamide riboside 1000mg twice daily). Group mean uric acid levels will be compared by paired t-test, with correction for multiple comparisons.
Effect of nicotinamide riboside on serum alanine aminotransferase levels | 9 days
  Comparison of group mean serum alanine aminotransferase levels at day 1 (baseline) vs. day 9 (while on nicotinamide riboside 1000mg twice daily). Group mean alanine aminotransferase levels will be compared by paired t-test, with correction for multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D O'Brien, MD, Principal Investigator — University of Washington; Rong Tian, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Airhart SE, Shireman LM, Risler LJ, Anderson GD, Nagana Gowda GA, Raftery D, Tian R, Shen DD, O'Brien KD. An open-label, non-randomized study of the pharmacokinetics of the nutritional supplement nicotinamide riboside (NR) and its effects on blood NAD+ levels in healthy volunteers. PLoS One. 2017 Dec 6;12(12):e0186459. doi: 10.1371/journal.pone.0186459. eCollection 2017. PMID 29211728